CLINICAL TRIAL: NCT04490070
Title: Caregiver Training: Evidence of Its Effectiveness for Cognitive and Functional Improvement in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Miriam Sanjuan, Principal Investigator, Universidad de Granada
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 545/CEIH/2018
Record Dates: First submitted 2020-07-23; First posted 2020-07-28 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Functional Ability; Cognitive Decline; Older Adults; Healthy Aging
Keywords: Older adults; Caregiver training program; Cognitive stimulation; Professional caregivers; Family caregivers
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Cognitive Stimulation — The caregiver training program consisted of applying the cognitive stimulation model of the CUIDA-2 program. This application included theoretical training made up of three modules: 1) person-centered care, 2) communication strategies, and 3) mediated cognitive stimulation strategies. The training was given in two group sessions of two hours each, plus 50 hours of individual practice, either on the job (in the case of professional caregivers) or in the home (in the case of family caregivers), in both cases supervised by psychologists who were experts in the program. In these individual practice hours, the caregivers were required to keep a weekly log. Here they had to plan in advance the activities that they were going to carry out with the older adult, and once they had taken place, they had to record how they were done and how the older adult had responded.

SUMMARY:
Due to demographic changes that have resulted in an aging population, the role of caregiver of an older adult has become very important in recent years. While numerous programs have been designed to lighten the caregiver's physical and emotional burden, fewer programs train caregivers to improve skills and level of independence in the person they care for. The objectives of this research study were to assess the benefits of a caregiver training program on the cognitive and functional status of older adults, as well as to compare the effects of this program according to type of caregiver (professional caregiver vs. family caregiver). Methods: The sample was composed of 160 older adults: a) 100 received care from caregivers who had taken the training program (treatment group), of which 60 were professional caregivers and 40 were family caregivers; and b) 60 received care from caregivers who had not taken the program (control group). In order to evaluate program effects on cognitive and functional status, we used both direct measures (MMSE, CAPE and EuroQol) and caregiver reports (Barthel and RMPBC).

ELIGIBILITY:
Inclusion Criteria:

* Older adults: age 65 or older, receiving care, no diagnosis of dementia, and their informed consent.

Exclusion Criteria:

-

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 160 (Actual)
Dates: Start 2015-12-10 (Actual); Primary Completion 2020-03-10 (Actual); Study Completion 2020-03-10 (Actual)

PRIMARY OUTCOMES:
Mini-Examen-Cognoscitivo (MEC), Spanish adaptation of the Mini-Mental-State-Examination (MMSE). | 9 months
  This screening instrument is widely used for detecting cognitive impairment. The final score ranges from 0 to 35 points and is often used as a global index and method for monitoring the evolution of cognitive functions in cognitive impairment and dementia. It has high internal consistency (α = 0.88), good test-retest reliability (0.64-1.00; p < 0.01) and good interjudge reliability (0.69-1.00; p < 0.01).
The Procedimiento de Evaluación Clifton para Ancianos - Cognitive Scale, a Spanish adaptation of the Clifton Assessment Procedure for the Elderly (CAPE). | 9 months
  In the present study, we used the cognitive assessment scale only, which includes one part on information and orientation and another part on mental ability. The final score ranges from 0 to 23 points and higher scores mean a better outcome. Its test-retest reliability falls between 0.79 and 0.90, and between 0.61 and 0.69, for the information and orientation scale and for the mental ability scale, respectively.
EuroQol | 9 months
  Generic measure of health-related quality of life. The individual rates his or her own state of health, first rating levels of severity by dimensions, and afterward a more general assessment using a 20-centimeter visual analog scale (VAS) that goes from 0 to 100. Scores range from 0 to 2 on each of the test scales, and higher scores mean a worse result.
Barthel Index | 9 months
  Evaluates the person's functional ability based on 10 items answered by the caregiver. Scores range from 0 to 100, with 0 being completely dependent and 100 completely independent. Its internal consistency presents an alpha coefficient between 0.86 and 0.92 and interjudge reliability between 0.84 and 0.97.
Revised Memory and Behavior Problem Checklist (RMBPC), in its Spanish version. | 9 months
  Evaluates problems in memory, behavior, and anxiety and depression. The caregiver indicates how often the person under her care has manifest each of the problems described during the past week (frequency scale) and the degree that this bothers or worries her (reaction scale). An alpha coefficient of 0.84 was found for the frequency scale, and 0.90 for the reaction scale.
Positive Aspects of Caregiving (PAC). | 9 months
  This 9-item instrument measures caregivers' satisfaction with providing care to the older adults. It consists of a 5-point Likert scale from 1 (disagree) to 5 (agree). Scores range from 9 to 45; higher scores indicate a more positive perception and gains from the caregiver experience. It presents good general reliability (Cronbach α = .89) and convergent validity (Cronbach α = .72).

CONTACTS AND LOCATIONS:
Overall Officials: Elena Navarro, Study Director — Universidad de Granada; Dolores Calero, Study Chair — Universidad de Granada; Miriam Sanjuán, Principal Investigator — Universidad de Granada
Locations (10):
- Spain (10):
  - Centro Residencial de Mayores "Entreálamos", Atarfe, Granada
  - Unidad de Estancia Diurna de Atarfe, Atarfe, Granada
  - Residencia de mayores María Zayas, Belicena, Granada
  - Centro Residencial Regina Mundi, Churriana de la Vega, Granada
  - Centro Residencial Geriatric XXI, Cúllar-Vega, Granada
  - Unidad de Estancia Diurna Ogíjares, Ogíjares, Granada
  - Unidad de Estancia Diurna Dr. Alejandro Otero, Pulianas, Granada
  - Centro Cívico Zaidín del Ayuntamiento de Granada, Granada
  - Centro Cívico Genil del Ayuntamiento de Granada, Granada
  - University of Granada, Granada

IPD SHARING:
Plan to Share IPD: No